CLINICAL TRIAL: NCT06497439
Title: Efficacy and Safety of Silfamin for Common Cold With or Without Sore Throat: Preliminary Study
Brief Title: Efficacy and Safety of Silfamin for Common Cold
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRSU.P.Dexa/06/20/14.04
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Common Cold; Sore-throat
Keywords: Common Cold; Sore-throat; Silfamin
MeSH Terms: conditions — Common Cold; Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silfamin (Experimental): 2 tablets of Silfamin 150 mg twice daily
  Interventions: Drug: Silfamin
- Placebo (Placebo Comparator): 2 tablets of Placebo twice daily
  Interventions: Drug: Placebo tablet of Silfamin

INTERVENTIONS:
Drug: Silfamin — 2 tablets of Silfamin 150 mg twice daily
  Other Names: Herbacold
  Arms: Silfamin
Drug: Placebo tablet of Silfamin — 2 tablets of Silfamin Placebo twice daily
  Arms: Placebo

SUMMARY:
This is a 2-arm, prospective, randomized, double-blind, placebo-controlled, and three-days-treatment clinical study comparing the efficacy and safety of Silfamin at a dose of 2 tablets@150 mg twice daily in subjects with common cold.

DETAILED DESCRIPTION:
There will be 2 groups of treatment; each group will consist of 30 subjects receiving the following regimens for three days:

Treatment I : 2 tablets of Silfamin 150 mg 2 times daily Treatment II : 2 tablets of Placebo 2 times daily

Eligible subjects will be evaluated for treatment efficacy at 0 hours (just before drug administration), 1 and 2 hours after the first dose. For the next doses, subject will perform a self-assessment for treatment efficacy at 1 and 2 hours after every dosing, and record it in subject's diary.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy (by anamnesis) men or women aged 18 to 60 years with mild or moderate common cold with or without sore throat (Common cold Score of 1 or 2)
* Willing to participate in the study by signing the informed consent

Exclusion Criteria:

* Body temperature of > 37.3˚C and/or refuse to follow health protocol for COVID-19
* Known hypersensitivity to herbal drugs containing Nigella sativa and/or Phaleria macrocarpa
* Pregnant or lactating women
* Have received any analgesic, anti-inflammatory or other common cold preparation within the past 24 hours
* Presence of vomiting or diarrhea within the past 24 hours and still ongoing at the start of study
* Severe illness, e.g. severe hypertension (> 160/100 mmHg)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Score of common cold and sore throat | 30 minutes, 60 minutes, 90 minutes, 2 hours, 1 day, 2 days, 3 days
  Score of common cold and sore throat measured at 0 hours (just before drug administration) for the first dose, 1 and 2 hours after every dosing
VAS score of sore throat | 30 minutes, 60 minutes, 90 minutes, 2 hours, 1 day, 2 days, 3 days
  VAS score of sore throat measured at 0 hours (just before drug administration), 1 and 2 hours after every dosing

SECONDARY OUTCOMES:
Adverse events | 1, 2, 3 days
  Number of adverse event, will be observed throughout the study conduct

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - IMERI Faculty of Medicine, University of Indonesia, Jakarta Pusat, Jakarta Special Capital Region
  - Makara UI Satellite Clinic, Depok, West Java